CLINICAL TRIAL: NCT00103194
Title: Phase II Trial of GW572016 in Patients With Recurrent Prostate Cancer as Evident by a Rising PSA
Brief Title: Lapatinib Ditosylate in Treating Patients With a Rising PSA Indicating Recurrent Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-01158; NCI-2014-01158 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); E5803 (Other: Eastern Cooperative Oncology Group (ECOG)); CDR0000409729; U10CA180820 (NIH); U10CA021115 (NIH); NCT02154373 (obsolete NCT alias)
Record Dates: First submitted 2005-02-07; First posted 2005-02-08 (Estimated); Results first posted 2012-04-13 (Estimated); Last update posted 2014-09-30 (Estimated); Status verified 2014-06

CONDITIONS: Recurrent Prostate Cancer; Stage I Prostate Cancer; Stage IIA Prostate Cancer; Stage IIB Prostate Cancer; Stage III Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Lapatinib; N-(3-chloro-4-((3-fluorobenzyl)oxy)phenyl-6-(5-((methylsulfonyl)ethyl)aminomethyl)-2-furyl)-4-quinazolinamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (lapatinib ditosylate) (Experimental): Patients receive lapatinib ditosylate PO daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: lapatinib ditosylate; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: lapatinib ditosylate — Given PO
  Other Names: GSK572016; GW-572016; GW2016; Lapatinib; Tykerb
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial studies how well lapatinib ditosylate works in treating patients with a rising prostate-specific antigen (PSA), a protein made by the prostate gland, indicating that prostate cancer has come back after previous treatment. Lapatinib ditosylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and may delay or prevent the progression of prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the percentage of patients with hormone sensitive prostate cancer who experience > 50% decline in serum PSA during treatment with GW572016 (lapatinib ditosylate).

SECONDARY OBJECTIVES:

I. To evaluate the duration of PSA decline. II. To characterize the change in PSA slope with GW572016. III. To characterize the safety and tolerability of GW572016 in this patient population.

IV. To estimate the time to progression (TTP) and progression-free survival at 2 years (from start of therapy).

V. To evaluate the correlation of epidermal growth factor receptor (EGFR) expression/signaling (from available prostate biopsy specimens or prostatectomy blocks) and its relationship to change in PSA in patients treated with GW572016.

OUTLINE:

Patients receive lapatinib ditosylate orally (PO) daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months if patient is < 2 years from study entry, every 6 months if patient is 2-5 years from study entry, or every year if patient is 5-10 years from study entry for 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of prostate cancer
* Previous treatment with definitive surgery or radiation therapy
* Prior salvage therapy (surgery, radiation, or other local ablative procedures) is allowed if the intent was for cure
* No evidence of metastatic disease on physical exam, computed tomography (CT) (magnetic resonance imaging [MRI]), and bone scan
* Prior neoadjuvant/adjuvant hormonal or chemotherapy and investigational agents are allowed if it was last used >= 1 year prior to enrollment (no prior vaccine/immunotherapy for prostate cancer will be allowed)
* No therapy modulating testosterone levels (such as luteinizing-hormone releasing-hormone agonists/antagonists and antiandrogens) is permitted within 1 year prior to enrollment; agents such as 5alpha-reductase inhibitors, ketoconazole, megestrol acetate, systemic steroids, or herbal supplements are not permitted at any time during the period that the PSA values are being collected
* Hormone-sensitive prostate cancer as evident by a serum total testosterone level > 150 ng/dL within 4 weeks prior to registration
* All patients must have evidence of biochemical progression as determined by a reference PSA value followed by 2 rising PSA values, each higher than the previous value, obtained at least 6 weeks apart; all of these PSA values must be obtained at the same reference lab, and all must be done within 6 months prior to enrollment
* The most recent of the PSA values must be greater than 0.4 ng/ml (after prostatectomy) or greater than 1.5 ng/ml (after radiation therapy) at time of enrollment; this measurement must be obtained within 6 months prior to enrollment
* PSA doubling time (PSADT) must be =< 365 days
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1
* Leukocytes >= 3000/mm^3
* Granulocytes >= 1500/mm^3
* Platelet count >= 100,000/mm^3
* Serum creatinine within normal institutional limits or creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Serum total bilirubin within normal institutional limits
* Serum alkaline phosphatase within normal institutional limits
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) and serum glutamic pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 2.5 x institutional upper limit of normal
* Cardiac ejection fraction within the institutional range of normal, as measured by echocardiogram or multi gated acquisition scan (MUGA) scan within 4 weeks prior to registration; note that baseline and on-treatment scans should be performed using the same modality and preferably at the same institution
* No unstable arrhythmias on electrocardiogram (ECG) are allowed (rate controlled, asymptomatic atrial fibrillation is allowed)
* No concomitant use of any medication classified as cytochrome P450 family 3, subfamily A, polypeptide 4 (CYP3A4) inducer or inhibitor; for patients previously treated with one of these prohibited medications, the prohibited agent needs to be discontinued, either 7 days, 14 days, or 6 months prior to the administration of the first dose of study medication
* Human immunodeficiency virus (HIV)-positive patients receiving combination anti-retroviral therapy are excluded from the study; appropriate studies will be undertaken in patients receiving combination anti-retroviral therapy when indicated
* Normal prothrombin time (PT)/international normalized ratio (INR) within 4 weeks prior to registration
* Able to swallow and retain oral medication
* Patients with gastrointestinal (GI) tract disease resulting in an inability to take oral medication, malabsorption syndrome, a requirement for intravenous (IV) alimentation, prior surgical procedures affecting absorption, uncontrolled inflammatory GI disease (e.g., Crohn's, ulcerative colitis) will not be eligible
* Sexually active males are strongly advised to use an accepted and effective method of contraception
* Patients may not be receiving any other investigational agents or receiving concurrent anticancer therapy
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to GW572016
* No uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* No other malignancies permitted within the past 5 years with the exception of non-melanoma skin cancer treated with curative intent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2005-09; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Liu, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (1):
- ECOG-ACRIN Cancer Research Group, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Liu G, Chen YH, Kolesar J, Huang W, Dipaola R, Pins M, Carducci M, Stein M, Bubley GJ, Wilding G. Eastern Cooperative Oncology Group Phase II Trial of lapatinib in men with biochemically relapsed, androgen dependent prostate cancer. Urol Oncol. 2013 Feb;31(2):211-8. doi: 10.1016/j.urolonc.2011.01.002. Epub 2011 Jul 23. PMID 21784672

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from ECOG member institutions between September 29, 2005 and July 5, 2006.
Groups:
- GW572016 (Lapatinib): GW572016 was administered at a dose of 1500 mg orally daily on an outpatient basis. Patients were advised to take GW572016 on an empty stomach (either 1 hour before or 1 hour after meals). GW572016 was administered continuously until disease progression or unacceptable toxicities. For the purposes of protocol evaluations, a cycle was defined as 28 days.
Period: Overall Study
Arm/Group | GW572016 (Lapatinib)
Started | 49
Treated | 49
Eligible | 35
Eligible and Treated | 35
Completed | 18
Not Completed | 31

BASELINE CHARACTERISTICS:
Arm/Group | GW572016 (Lapatinib)
Number analyzed (Participants) | 35
Age, Continuous [Median (Full Range); unit: years] — Age of eligible patients who began treatment.
  years | 65 [48 to 81]
Sex: Female, Male [Count of Participants; unit: Participants] — Gender of eligible patients who began treatment.
  Participants
    Female | 0
    Male | 35

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With PSA Response, Defined as a 50% or Greater Decline in the Serum PSA Level
Description: PSA response is defined as either complete response (CR) or partial response (PR) observed at any time during the entire measurement time period.
  CR: In patients treated with prior radical prostatectomy, a PSA < 0.2 ng/mL confirmed by a repeat PSA at least one month apart was considered a complete biochemical response. In patients treated with radiation therapy only, a PSA < 1 ng/mL on three separate occasions taken at least one month apart was considered a complete biochemical response.
  PR: A reduction in PSA by > 50% from baseline, confirmed by repeat PSA 1 month later.
Time Frame: Assessed every cycle while on treatment; after being off-treatment, assessed every 3 months for 2 years, then every 6 months for 3 years, then annually for 5 years
Population: Eligible patients who started protocol treatment
Measure: Number; unit: participants
Arm/Group | GW572016 (Lapatinib)
Number analyzed (Participants) | 35
participants
  Response | 0
  Stable Disease | 28
  Progression | 4
  Unevaluable | 3
Statistical Analysis 1: Comparison: GW572016 (Lapatinib); Test type: Superiority or Other; PSA response rate = 0, 90% CI 2-sided [0 to 8.2]

2. Secondary Outcome: The Change in PSA Slope With GW572016 (Lapatinib)
Description: PSA was evaluated every cycle while on treatment. PSA test results show the level of PSA detected in the blood. These results were reported as nanograms of PSA per milliliter (ng/mL) of blood. PSA slope is the change in PSA level over time. A sharp rise in the PSA level raises the suspicion of cancer and may indicate a fast-growing cancer.
Time Frame: Assessed every cycle while on treatment; after being off-treatment, assessed every 3 months for 2 years, then every 6 months for 3 years, then annually, for 5 years
Population: One patient who withdrew from study after receiving 4 days of treatment and did not have any follow-up PSA measurements was excluded from this analysis, so the number of participants analyzed is 34.
Measure: Mean (Standard Error); unit: log (PSA)/month
Arm/Group | GW572016 (Lapatinib)
Number analyzed (Participants) | 34
log (PSA)/month
  Pre-treatment PSA slope | 0.19 (0.019)
  Post-treatment PSA slope | 0.13 (0.017)
Statistical Analysis 1: Comparison: GW572016 (Lapatinib); Test type: Superiority or Other; p = 0.006, Mixed Models Analysis; The analysis is testing the null hypothesis that there is no difference between the pre-treatment and post-treatment PSA slopes

3. Secondary Outcome: Progression-free Survival Rate at 2 Years
Description: Proportion of patients who are living with a disease that does not get worse at 2 years from registration based on Kaplan-Meier method.
Time Frame: as for outcome 1
Population: Eligible patients who started treatment.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | GW572016 (Lapatinib)
Number analyzed (Participants) | 35
percentage of participants | 16.0 [6.5 to 29.1]

4. Secondary Outcome: Relationship Between Progression-free Survival and EGFR Expression Levels
Description: The association between EGFR (epidermal growth factor receptor) expression levels and the length of time during and after treatment in which a patient is living with a disease that does not get worse.
Time Frame: as for outcome 1
Population: Eligible patients who started treatment.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | GW572016 (Lapatinib)
Number analyzed (Participants) | 35
months
  High EGFR | 17.4 [4.7 to 20.9]
  Low EGFR | 6.0 [3.0 to 12.4]

ADVERSE EVENTS:
Time Frame: Assessed every 4 weeks while on treatment and for 30 days after the end of treatment.
Arm/Group | GW572016 (Lapatinib)
Serious Adverse Events (participants affected / at risk) | 4/49
Other Adverse Events (participants affected / at risk) | 46/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GW572016 (Lapatinib) (N=49)
Fatigue (General disorders) | 1
AST Increased (Investigations) | 1
Bilirubin Increased (Investigations) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GW572016 (Lapatinib) (N=49)
Anemia (Blood and lymphatic system disorders) | 4
Fatigue (General disorders) | 23
Insomnia (Psychiatric disorders) | 4
Dry Skin (Skin and subcutaneous tissue disorders) | 6
Flushing (Vascular disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 3
Nail Changes (Skin and subcutaneous tissue disorders) | 6
Pruritus/Itching (Skin and subcutaneous tissue disorders) | 6
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 9
Rash: Acne/Acneiform (Skin and subcutaneous tissue disorders) | 35
Skin- Other (Skin and subcutaneous tissue disorders) | 5
Anorexia (Metabolism and nutrition disorders) | 4
Constipation (Gastrointestinal disorders) | 3
Diarrhea w/o Prior Colostomy (Gastrointestinal disorders) | 34
Flatulence (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 3
Nose, Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 3
ALT Increased (Investigations) | 9
AST Increased (Investigations) | 7
Bilirubin Increased (Investigations) | 9
Hyperglycemia (Metabolism and nutrition disorders) | 4
Neuropathy-Sensory (Nervous system disorders) | 4
Abdominal Pain (Gastrointestinal disorders) | 5
Headache (Nervous system disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less